CLINICAL TRIAL: NCT01637844
Title: Telbivudine in the Third Trimester of Pregnancy to Prevent Mother-to-infant Transmission of HBV
Brief Title: Telbivudine Therapy in HBeAg-positive Pregnant Women to Prevent Mother-to-infant Transmission of HBV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yi-Hua Zhou (Other)
Collaborators: Taixing People's Hospital (Other); Fourth People's Hospital of Zhenjiang, China (Other); Wuxi Maternal and Child Health Hospital (Unknown); The First People's Hospital of Kunshan (Other)
Responsible Party: Sponsor-Investigator, Yi-Hua Zhou, Professor of Infectious Diseases, Chair of Experimental Medicine, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012019
Record Dates: First submitted 2012-07-04; First posted 2012-07-11 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: HBV
Keywords: Pregnant women; HBsAg positive; HBeAg positive; Telbivudine
MeSH Terms: interventions — Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telbivudine (Experimental): HBsAg- and HBeAg-positive pregnant women at 28-32 weeks of gestation start to orally take telbivudine (600 mg/day) until 4 weeks after delivery. Newborn infants receive standard immunoprophylaxis.
  Interventions: Drug: Telbivudine
- Control (No Intervention): Infants of HBsAg- and HBeAg-positive women who are not treated with telbivudine and any other antiviral agents serve as controls. The infants are administered standard immunoprophylaxis against mother-to-infant transmission of HBV, 100-200 IU hepatitis B immunoglobulin (HBIG) within 12 hours after birth and three doses hepatitis B vaccine at 0, 1 and 6-month schedule.

INTERVENTIONS:
Drug: Telbivudine — HBsAg- and HBeAg-positive pregnant women at 28-32 weeks of gestation are given with telbivudine (oral 600 mg/day) until 4 weeks after delivery. Newborn infants are administered 100-200 IU HBIG within 12 hours after birth and vaccinated against hepatitis B with yeast recombinant hepatitis B vaccine (10 µg) at 0, 1, and 6-month schedule. HBV DNA and ALT levels are measured before the use of telbivudine, at delivery, and 1-2 months after stopping the drug. HBV serological markers, including HBsAg, anti-HBs, and anti-HBc, HBeAg and anti-HBe are tested in infants at age of 7-12 months.
  Other Names: Anti-HBV therapy during pregnancy
  Arms: Telbivudine

SUMMARY:
Infants of hepatitis B virus (HBV)-infected mothers with positive hepatitis B e antigen (HBeAg) have an increased risk of becoming infected with HBV. This study will determine whether telbivudine among both hepatitis B surface antigen (HBsAg) and HBeAg positive pregnant women during the third trimester, in addition to standard immunoprophylaxis in infants, will be more effective than standard immunoprophylaxis alone at preventing HBV infections in these infants.

DETAILED DESCRIPTION:
Infants of HBV-infected mothers with positive HBeAg have an increased risk of becoming infected with HBV. Standard immunoprophylaxis against mother-to-infant transmission of HBV includes administration of hepatitis B immunoglobulin (HBIG) and hepatitis B vaccine; however, approximately 5-15% of the infants are not protected despite having received these preventive measures. It is reported that antiviral prophylaxis among HBV-infected pregnant women can reduce mother-to-infant transmission of HBV. However, more research is needed to obtain the definite conclusion. This study will determine whether telbivudine among HBsAg- and HBeAg-positive pregnant women during the third trimester, in addition to standard immunoprophylaxis in infants, will be more effective than standard immunoprophylaxis alone at preventing HBV infections in these infants.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at 28-32 weeks of gestation
* both HBsAg and HBeAg positive
* good compliance

Exclusion Criteria:

* Coinfection of HAV, HCV, HEV, HIV, and STD
* With history of antiviral treatment against HBV
* With chronic disease, such as heart and kidney disease, asthma, diabetes, hyperthyroidism, severe anemia, bleeding disease, autoimmune diseases
* With threatened miscarriage or relevant treatment during the pregnancy
* With pregnant complications such as pregnancy hypertension, preeclampsia, etc
* With history of fetal deformity, or fetal deformity detected by ultrasound examination
* With ALT >10 times upper limit, or total bilirubin >3 times upper limit, of normal value

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 335 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
HBV serologic markers and alanine transaminase (ALT) levels in infants | 10 months after birth
  HBsAg and HBeAg are tested in umbilical blood and peripheral blood collected at the age of 10 months respectively. ALT is measured at 10 months old.

SECONDARY OUTCOMES:
HBV DNA quantification and ALT levels in mothers | Up to 10 months postpartum
  HBV DNA and ALT levels in the pregnant women are measured before taking telbivudine, at birth, 1-2 months after stopping the drug, and 10 months postpartum.
Women and infants with adverse events | Up to 10 months after delivery/birth
  Adverse events in pregnant women during pregnancy, complications at delivery and postpartum, Apgar score, newborn infant deformity, infant growth and development will be recorded during the study period (up to 10 months after delivery/birth).

CONTACTS AND LOCATIONS:
Overall Officials: Yali Hu, MD, PhD, Study Director — Nanjing Drum Tower Hospital, Nanjing University Medical School
Locations (3):
- China (3):
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Taixing People's Hospital, Taishing, Jiangsu
  - Zhenjiang Fourth People's Hospital, Zhenjiang, Jiangsu

REFERENCES:
- [Background] Han GR, Cao MK, Zhao W, Jiang HX, Wang CM, Bai SF, Yue X, Wang GJ, Tang X, Fang ZX. A prospective and open-label study for the efficacy and safety of telbivudine in pregnancy for the prevention of perinatal transmission of hepatitis B virus infection. J Hepatol. 2011 Dec;55(6):1215-21. doi: 10.1016/j.jhep.2011.02.032. Epub 2011 Apr 15. PMID 21703206
- [Background] Pan CQ, Han GR, Jiang HX, Zhao W, Cao MK, Wang CM, Yue X, Wang GJ. Telbivudine prevents vertical transmission from HBeAg-positive women with chronic hepatitis B. Clin Gastroenterol Hepatol. 2012 May;10(5):520-6. doi: 10.1016/j.cgh.2012.01.019. Epub 2012 Feb 14. PMID 22343511
- [Derived] Hu Y, Xu C, Xu B, Hu L, Liu Q, Chen J, Liu J, Liu L, Yang J, Chen T, Wen J, Jiang N, Zhang Y, Cao M, Feng J, Lin X, Wang Z, Xu B, Zhou YH. Safety and efficacy of telbivudine in late pregnancy to prevent mother-to-child transmission of hepatitis B virus: A multicenter prospective cohort study. J Viral Hepat. 2018 Apr;25(4):429-437. doi: 10.1111/jvh.12834. Epub 2017 Dec 26. PMID 29193547